CLINICAL TRIAL: NCT05052372
Title: Biomarker Research Study for Patients With FGFR-Mutant Bladder Cancer Receiving Erdafitinib
Status: Terminated | Type: Observational
Why Stopped: Sponsor request to terminate study due to enrollment numbers
Sponsor: xCures (Industry)
Responsible Party: Sponsor
Other Study IDs: TYRA-001-BC-2021
Record Dates: First submitted 2021-09-10; First posted 2021-09-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2021-09

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Transitional Cell Carcinoma; Platinum-Resistant Urothelial Carcinoma; Bladder Urothelial Carcinoma; FGFR Mutation; FGFR2 Gene Mutation; FGFR3 Gene Mutation; FGFR2 Amplification; Locally Advanced Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Refractory Bladder Carcinoma; Refractory Bladder Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — erdafitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liquid biopsies (blood and urine) will be collected at two or three timepoints per each patient approximately within a 2 to 15 month timeframe.
  3 x 10 mL ctDNA whole blood collection
  1 x 5 mL Random Urine collection
  DNA from blood plasma and urine will be isolated and tumor DNA will be purified.
  Samples will be stored securely and may be kept for up to 5 years after the last subject completes the study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Balversa — BALVERSA® is a prescription medicine used to treat adults with bladder cancer (urothelial cancer) that has spread or cannot be removed by surgery

SUMMARY:
Bladder cancers are associated with genetic mutations that are present in the patient's bladder or urothelium, the lining of the lower urinary tract. Fibroblast growth factor (FGFR) alterations are present in approximately one in five patients with recurrent and refractory bladder cancer.

This study will collect biomarker data from subjects receiving erdafitinib to further investigate the relationship between treatment with erdafitinib and clinical response, progression, and/or genetic alterations.

DETAILED DESCRIPTION:
The purpose of this study is to collect biomarker data from subjects receiving standard of care erdafitinib to further investigate the relationship between treatment with erdafitinib and clinical response, progression, and/or genetic alterations in cell free tumor DNA (cfDNA) from blood and urine samples.

In this study, next generation sequencing of cfDNA isolated from blood and urine will be performed by Resolution Bioscience. Blood-based cfDNA amplification and analysis is done by a CLIA-approved assay and the results of which will thus be available to physicians and patients. Urine-based cfDNA analysis from Resolution Bioscience is not yet approved and results will only be communicated if an actionable finding is identified that is not present on the blood-based test. Samples will be collected at the patients homes by a qualified phlebotomist.

xCures may provide the treating physician and the subject the biomarker results from blood-based cfDNA tests. Because the testing of urine DNA is experimental and done solely for research, those results will not be shared unless there is an important finding known to be relevant to the subject's medical care at the time of the study. The genetic tests are not approved for bladder cancer, so the information generated from biomarker research studies is preliminary in nature. Therefore, the significance and scientific validity of the results are undetermined. xCures and/or Tyra may additionally share data with the treating physician and researchers for the purposes of publication.

Patients co-enroll in an observational research study (XCELSIOR, NCT03793088) and consent to provide xCures right of access to their full medical records under HIPAA.

Patient clinical data is structured and centralized by xCures in a 21 CFR Part 11-compliant REDCap Cloud database in Case Report Forms (CRFs). The CRFs are a set of electronic forms for each patient that provides a record of clinical data generated according to the protocol. Data is abstracted directly from medical records generated in the standard practice of medicine.

xCures will request medical records directly from treating institutions and from other providers (commercial next generation sequencing providers, for example) and will work with treating physicians to ensure the completeness and accuracy of CRF content based on electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of locally advanced or metastatic bladder cancer
* Documented proof of an FGFR alteration according to a CLIA-based test
* Subjects who are receiving or will receive erdafitinib as their standard medical therapy as a monotherapy or in combination
* Age greater than or equal to 18 years.
* Subject is a resident of or seeking care in the United States
* Able and willing to provide informed consent to this biomarker study
* Informed consent obtained for the XCELSIOR longitudinal outcomes registry (NCT03793088).

Exclusion Criteria:

* Subjects younger than 18 years of age
* Subjects unwilling or unable to provide informed consent
* Subjects that are not receiving treatment in the United States or US Territories

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the United States with a diagnosis of locally advanced or metastatic bladder cancer (TCC/UC) may be screened for this study. In order to enroll on the study, subjects must have documented proof of an FGFR alteration according to a CLIA-based test with planned treatment with erdafitinib, or currently undergoing treatment with erdafitinib.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Relationship between treatment with erdafitinib and clinical response | Time to progression will vary for each patient. We expect most patients to progress on erdafitinib within 2 to 15 months from baseline
  Specimen collection will be performed at the following timepoints to assess clinical response while being treated with erdafitinib:
  1. Baseline (prior to or within 7 days of starting erdafitinib)
  2. Suspicion of progression (optional)
  3. Post-progression

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. George, MD, Principal Investigator — Duke Health
Locations (1):
- xCures Virtual Site, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Facchinetti F, Hollebecque A, Bahleda R, Loriot Y, Olaussen KA, Massard C, Friboulet L. Facts and New Hopes on Selective FGFR Inhibitors in Solid Tumors. Clin Cancer Res. 2020 Feb 15;26(4):764-774. doi: 10.1158/1078-0432.CCR-19-2035. Epub 2019 Oct 4. PMID 31585937